CLINICAL TRIAL: NCT04334239
Title: Wirksamkeit Der Versorgung in Onkologischen Zentren
Brief Title: Effectiveness of Care in Certified Cancer Centres in Germany
Acronym: WiZen
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Tumorzentrum Regensburg, Institut für Qualitätssicherung und Versorgungsforschung, Universität Regensburg (Unknown); Arbeitsgemeinschaft Deutscher Tumorzenten e.V., ADT (Unknown); Wissenschaftliches Institut der AOK (WIdO) (Unknown)
Responsible Party: Principal Investigator, Jochen Schmitt., Prof. Dr. med. Jochen Schmitt, MPH, Technische Universität Dresden
Other Study IDs: 01VSF17020
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer; Breast Cancer; Ovarian Cancer; Cervix Cancer; Endometrial Cancer; Bronchial Cancer; Prostate Cancer; Head and Neck Tumor; CNS Tumor; Pancreatic Cancer
Keywords: quality of treatment; institution of treatment; certification; cancer centres; quality of care; treatment outcome; health services research
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Carcinoma, Bronchogenic; Prostatic Neoplasms; Head and Neck Neoplasms; Central Nervous System Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Cancer patients who have undergone substantial parts of inpatient treatment in a certified cancer centre.
  Interventions: Other: Oncological certification
- Control: Cancer patients who have not undergone inpatient treatment in a certified cancer centre.

INTERVENTIONS:
Other: Oncological certification — Oncological certification encompasses a variety of criteria such as treatment according to the clinical guidelines, staffing, technical infrastructure, minimum caseloads, and multidisciplinary care.
  Groups: Intervention

SUMMARY:
Assessment of the effectiveness of care in certified cancer centres for eight cancer entities via a retrospective cohort study based on secondary data from statutory health insurance funds and population-based clinical cancer registries.

DETAILED DESCRIPTION:
Cancer constitutes the second most frequent cause of death in Germany. To maintain a high quality of treatment, the national cancer plan aims at a unified certification of cancer centres.

The project "Wirksamkeit der Versorgung in onkologischen Zentren" (WiZen) investigates effects of treatments in certified cancer centres across large populations and different cancer entities in comparison to hospitals that do not hold a certificate.

WiZen is a retrospective comparative cohort study that analyzes incident cases of eight types of cancer diagnosed within 2009-2017 based on nationwide health insurance data provided by WIdO (the AOK research institute) and data from regional clinical cancer registries (CCR) for the period 2006-2017. These eight types of cancer are colorectal cancer, pancreatic cancer, breast cancer, gynecologic tumors, lung cancer, prostate cancer, head and neck tumors and neuro-oncological tumors.

ELIGIBILITY:
Inclusion Criteria:

* first hospitalization due to diagnosis of colorectal cancer, pancreatic cancer, breast cancer, gynecologic tumors, lung cancer, prostate cancer, head and neck tumors, or neuro-oncological tumors 2009-2017 [WIdO]
* hospitalization due to primary diagnosis of colorectal cancer, pancreatic cancer, breast cancer, gynecologic tumors, lung cancer, prostate cancer, head and neck tumors, or neuro-oncological tumors 2006-2017 [CCR]

Exclusion Criteria:

* prevalent diagnosis of colorectal cancer, pancreatic cancer, breast cancer, gynecologic tumors, lung cancer, prostate cancer, head and neck tumors, or neuro-oncological tumors 2006-2017
* exception: outpatient cancer diagnosis up to 12 months prior to first hospitalization is not regarded as prevalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: German residents with continuous insurance of one of the AOK funds 2006-2017 and patients recorded in one of the participating cancer registries Dresden, Erfurt, Regensburg and Berlin-Brandenburg 2006-2017
Sampling Method: Non-Probability Sample
Enrollment: 670000 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | first hospitalization (starting from 01/01/2009 [WIdO] or 01/01/2006 [CCR]), up to 31/12/2017
  Survival after first hospitalization due to cancer
1- and 5-year survival | first hospitalization (starting from 01/01/2009 [WIdO] or 01/01/2006 [CCR]) with 1 or 5-year follow-up, respectively
  1- and 5-year survival after first hospitalization due to cancer
30-day mortality | first hospitalization (starting from 01/01/2009 [WIdO] or 01/01/2006 [CCR]) with 30 days follow-up
  30-day mortality after first hospitalization due to cancer

SECONDARY OUTCOMES:
2-, 3-, 4-year survival | first hospitalization (starting from 01/01/2009 [WIdO] or 01/01/2006 [CCR]) with 2,3, or 4-year follow-up, respectively
  2-, 3-, 4-year survival after first hospitalization due to cancer
Recurrence-free survival | cancer diagnosis (starting from 01/01/2009 [WIdO] or 01/01/2006 [CCR]), up to 31/12/2017
  Recurrence-free survival after cancer diagnosis
Cumulative recurrence rate | cancer diagnosis (starting from 01/01/2009 [WIdO] or 01/01/2006 [CCR]), up to 31/12/2017
  Cumulative recurrence rate after cancer diagnosis
Complications due to surgery | date of initial cancer surgery with entity-specific follow-up
  Complications due to cancer surgery
Successive resection | second resection within three months of initial cancer surgery
  Second resection due to cancer
Entity-specific outcomes defined by clinical experts | 2009-2017 [CCR] or 2006-2017 [WIdO]
  1. Fractions of entity-specific surgery techniques
  2. For head-neck-tumours: aspiration pneumonia due to swallowing dysfunctions
Fraction of patients | 2009-2017
  Fraction of patients in certified centres and in non-certified hospitals over time
Regional differences | 2009-2017
  Differences across outcomes in different counties or federal states
Differences in patient characteristics | 2009-2017 [CCR] or 2006-2017 [WIdO]
  Differences in demographic characteristics, disease severity and risk factors across certified centres/non-certified hospitals
Pathways of treatment | 2009-2017
  Patient's treatment pathways among general practitioners, specialists, and hospitals w.r.t. certification
Severity Levels in insurance data | 2009-2017
  Deduction of cancer severity levels through linkage of health insurance and cancer registry data

CONTACTS AND LOCATIONS:
Locations (1):
- Technische Universität Dresden, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Hansinger J, Schoffer O, Volkel V, Gerken M, Wimberger P, Bierbaum V, Bobeth C, Rossler M, Droge P, Ruhnke T, Gunster C, Kleihues-van Tol K, Link T, Kast K, Papathemelis T, Ortmann O, Schmitt J, Klinkhammer-Schalke M. Comparison of survival in ovarian cancer patients following treatment in certified gynecologic oncology centers and non-certified hospitals: a German retrospective cohort study (WiZen). J Ovarian Res. 2025 Nov 4;18(1):238. doi: 10.1186/s13048-025-01843-8. PMID 41188998
- [Derived] Roessler M, Schmitt J, Bobeth C, Gerken M, Kleihues-van Tol K, Reissfelder C, Rau BM, Distler M, Piso P, Gunster C, Klinkhammer-Schalke M, Schoffer O, Bierbaum V. Is treatment in certified cancer centers related to better survival in patients with pancreatic cancer? Evidence from a large German cohort study. BMC Cancer. 2022 Jun 7;22(1):621. doi: 10.1186/s12885-022-09731-w. PMID 35672675